CLINICAL TRIAL: NCT01367158
Title: Phase 2, Observer-Blind, Controlled, Randomized, Multi-Center Extension Study to Evaluate Safety, Tolerability and Immunogenicity of a Third Dose of One of Four Different Formulations of rMenB + MenACWY in Adolescents Who Previously Received the Same Study Vaccines
Brief Title: Safety, Tolerability and Immunogenicity of a Third Dose of One of Four Different Formulations of rMenB + MenACWY Combination Vaccine in Adolescents Who Previously Received the Same Study Vaccines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V102_02E1
Record Dates: First submitted 2011-06-03; First posted 2011-06-06 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal disease; vaccines; adolescents; prevention; Meningitis
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Meningitis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (11):
- 3ABCWY (Experimental): Two doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine plus one dose of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine in previous study and one dose of the same in current study
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine
- 2ABCWY (Experimental): Two doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine plus one dose of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine in previous study and one dose of Tdap in current study
  Interventions: Biological: Tdap
- 3ABx2CWY (Experimental): two doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine plus Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine in previous study and one dose of the same in current study
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine
- 2ABx2CWY (Experimental): two doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine plus one dose of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine in previous study and one dose of Tdap in current study
  Interventions: Biological: Tdap
- 3ABCWY+OMV (Experimental): Two doses Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine plus outer membrane vesicles (OMV) in previous study and one dose of the same in current study
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine
- 2ABCWY+OMV (Experimental): Two doses Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine plus outer membrane vesicles (OMV) in previous study and one dose of Tdap in current study
  Interventions: Biological: Tdap
- 3ABCWYqOMV (Experimental): Two doses of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine plus one quarter dose of outer membrane vesicles (qOMV) in previous study and one dose of the same in current study
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine
- 2ABCWYqOMV (Experimental): Two doses of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine plus one quarter dose of outer membrane vesicles (qOMV) in previous study and one dose of Tdap in current study
  Interventions: Biological: Tdap
- 3B (Active Comparator): Two doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine in previous study and one dose of the same in current study
  Interventions: Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- 2B (Active Comparator): Two doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine in previous study and one dose of Tdap in current study
  Interventions: Biological: Tdap
- 1ACWY (Active Comparator): One dose of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine followed by one dose of placebo and one dose of Tdap in current study
  Interventions: Biological: Tdap

INTERVENTIONS:
Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant vaccine — The lyophilized Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine reconstituted with one dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
  Arms: 3ABCWY; 3ABCWY+OMV; 3ABCWYqOMV; 3ABx2CWY
Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine — Liquid Meningococcal (group B) multicomponent recombinant adsorbed vaccine
  Arms: 3B
Biological: Tdap — Sterile liquid suspension of tetanus and diphtheria toxoids and acellular pertussis components intended for intramuscular injection
  Arms: 1ACWY; 2ABCWY; 2ABCWY+OMV; 2ABCWYqOMV; 2ABx2CWY; 2B

SUMMARY:
This study will evaluate safety, tolerability, and immunogenicity of a booster dose of a meningococcal vaccine formulation in adolescents.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to be enrolled into this study were male or female who completed study V102_02 (primary study), and:

1. who were 11 to 18 years at the time of enrollment in primary study;
2. who had given their written consent at the time of enrollment;
3. who were available for all the visits scheduled in the study (ie, not planning to leave the area before the end of the study period);
4. who were in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

1. History of any meningococcal vaccine administration;
2. Current or previous, confirmed or suspected disease caused by N meningitidis;
3. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N meningitidis infection within 60 days of enrollment;
4. Significant acute or chronic infection within the previous 7 days or fever (defined as temperature >38°C) within the previous 3 days;
5. Antibiotics within 7 days prior to enrollment or blood draw;
6. Pregnancy or nursing (breastfeeding) mothers;
7. Females of childbearing age who had not used or did not plan to use acceptable birth control measures, for the duration of the study. Oral, injected or implanted hormonal contraceptive, barrier methods (condom or diaphragm with spermicide); intrauterine device or sexual abstinence was considered acceptable forms of birth control. If sexually active the subject must have been using one of the accepted birth control methods at least two months prior to study entry;
8. Any serious chronic or progressive disease (eg, neoplasm, diabetes, cardiac disease, hepatic disease, progressive neurological disease or seizure disorder; autoimmune disease, human immunodeficiency virus infection or acquired immunodeficiency syndrome, blood dyscrasias, bleeding diathesis, signs of cardiac or renal failure or severe malnutrition).
9. Known or suspected impairment/alteration of the immune system, immunosuppressive therapy, including use of corticosteroids in immunosuppressive doses or chronic use of inhaled high-potency corticosteroids or immunostimulants within the previous 60 days. Use of topical corticosteroids administered during the study in limited areas (ie, eczema on knees or face or elbows) of the body was allowed;
10. Receipt of blood, blood products and/or plasma derivatives, or a parenteral immunoglobulin preparation within the previous 90 days;
11. History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component;
12. Individuals who received any other vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study or who were planning to receive any vaccine within 4 weeks from the study vaccines.
13. Individuals participating in any clinical trial with another investigational product 30 days prior to first study visit or had intent to participate in another clinical study at any time during the conduct of this study.
14. Individuals who were part of study personnel or close family members conducting this study.
15. Individuals with medical history or any illness that, in the opinion of the investigator, might interfere with the results of the study or posed additional risk to the subjects due to participation in the study.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 440 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (7):
- Chile (2):
  - CESFAM Gabriela Mistral:, Aurora de Chile 9872 - San Ramón, Saniago
  - Pontificia Universidad Catolica de Chile, Marcoleta 350, Santiago Metropolitan
- Colombia (3):
  - CAFAM, Avenida Carrera 68# 90-88 Piso 4, Bogota D.C.
  - Centro de Investigacion CafeSalud Medicina Prepagada, Carrera 14 No. 94-49 PisoSexto, Bogota D.C.
  - CAIMED, Carrera, Bogota D.C.
- Panama (2):
  - Indicasat:, Clayton, Ciudad Del Saber Edificio 219, Panama City
  - Health Research International: Centro Especializado san Fernando, Piso Numero 5, Consultorio 12; Via Espana, Las Sabanas,, Panama City

REFERENCES:
- [Derived] Saez-Llorens X, Aguilera Vaca DC, Abarca K, Maho E, Han L, Smolenov I, Dull P. Persistence of Meningococcal Antibodies and Response to a Third Dose After a Two-dose Vaccination Series with Investigational MenABCWY Vaccine Formulations in Adolescents. Pediatr Infect Dis J. 2015 Oct;34(10):e264-78. doi: 10.1097/INF.0000000000000822. PMID 26135245

RESULTS

PARTICIPANT FLOW:
Groups:
- 3ABCWY: Two doses of MenABCWY vaccine (no outer membrane vesicle {OMV}) in the primary study and one dose of the same vaccine in the current study
- 2ABCWY: Two doses of MenABCWY vaccine (no OMV) in the primary study and one dose of Tdap in the current study
- 3ABx2CWY: Two doses of MenABx2CWY vaccine in the primary study and one dose of the same vaccine in the current study
- 2ABx2CWY: Two doses of MenABx2CWY vaccine in the primary study and one dose of Tdap in the current study
- 3ABCWY+OMV: Two doses MenABCWY+OMV vaccine in the primary study and one dose of the same vaccine in the current study
- 2ABCWY+OMV: Two doses MenABCWY+OMV vaccine in the primary study and one dose of Tdap in the current study
- 3ABCWYqOMV: Two doses of MenABCWY+1/4OMV vaccine in the primary study and one dose of the same vaccine in the current study
- 2ABCWYqOMV: Two doses of MenABCWY+1/4OMV vaccine in the primary study and one dose of Tdap in the current study
- 3 B: Two doses of rMenB vaccine in the primary study and one dose of the same vaccine in the current study
- 2 B: Two doses of rMenB vaccine in the primary study and one dose of Tdap in the current study
- 1ACWY: One dose of MenACWY vaccine followed by one dose of placebo in the primary study and one dose of Tdap in the current study
Period: Overall Study
Arm/Group | 3ABCWY | 2ABCWY | 3ABx2CWY | 2ABx2CWY | 3ABCWY+OMV | 2ABCWY+OMV | 3ABCWYqOMV | 2ABCWYqOMV | 3 B | 2 B | 1ACWY
Started | 25 | 49 | 24 | 49 | 25 | 48 | 25 | 49 | 23 | 50 | 73
Completed | 25 | 46 | 23 | 48 | 23 | 46 | 25 | 47 | 23 | 50 | 72
Not Completed | 0 | 3 | 1 | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 1
Not completed — Withdrew consent | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3ABCWY | 2ABCWY | 3ABx2CWY | 2ABx2CWY | 3ABCWY+OMV | 2ABCWY+OMV | 3ABCWYqOMV | 2ABCWYqOMV | 3 B | 2 B | 1ACWY | Total
Number analyzed (Participants) | 25 | 49 | 24 | 49 | 25 | 48 | 25 | 49 | 23 | 50 | 73 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (2.2) | 14.2 (2.0) | 14.4 (2.1) | 14.4 (2.1) | 14.9 (2.6) | 14.2 (2.1) | 14.3 (2.0) | 14.4 (2.1) | 14.8 (2.5) | 15.0 (2.0) | 14.8 (2.1) | 14.5 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 29 | 14 | 27 | 12 | 26 | 14 | 19 | 11 | 25 | 39 | 232
  Male | 9 | 20 | 10 | 22 | 13 | 22 | 11 | 30 | 12 | 25 | 34 | 208

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With hSBA ≥1:8 Against Serogroups A, C, W and Y at One Month After the Third Vaccination With Either One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Description: Antibody response was measured as the percentage of subjects with human serum bactericidal assay (hSBA) titers ≥1:8 and associated 95% CI, directed against to N meningitidis serogroups A, C, W, and Y at 6 months following first vaccine during the parent study NCT01210885 and one month after third vaccination (Month 7).
Time Frame: At month 6 and month 7
Population: Analysis was done by Modified Intention-To-Treat (MITT) Month 7 Set. MITT is defined as all subjects in the enrolled set who received a study vaccination at Month 6 and provided one evaluable serum sample at Month 7.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- 3 B: Two doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine in previous study and one dose of the same in current study
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 72
Percentages of subjects
  Ser. A - month 6 (n=23,24,24,25,23,69) | 52 [31 to 73] | 79 [58 to 93] | 75 [53 to 90] | 68 [46 to 85] | 35 [16 to 57] | 55 [43 to 67]
  Ser. A - month 7 (n=24,24,21,25,22,71) | 100 [86 to 100] | 100 [86 to 100] | 100 [84 to 100] | 100 [86 to 100] | 91 [71 to 99] | 58 [45 to 69]
  Ser. C - month 6 (n=22,24,24,24,21,70) | 100 [85 to 100] | 96 [79 to 100] | 100 [86 to 100] | 100 [86 to 100] | 33 [15 to 57] | 76 [64 to 85]
  Ser. C - month 7 (n=23,24,23,25,22,72) | 100 [85 to 100] | 100 [86 to 100] | 100 [85 to 100] | 100 [86 to 100] | 73 [50 to 89] | 68 [56 to 79]
  Ser. W - month 6 (n=24,24,25,24,22,69) | 100 [86 to 100] | 96 [79 to 100] | 100 [86 to 100] | 100 [86 to 100] | 55 [32 to 76] | 97 [90 to 100]
  Ser. W - month 7 (n=23,24,21,25,21,72) | 100 [85 to 100] | 100 [86 to 100] | 100 [84 to 100] | 100 [86 to 100] | 90 [70 to 99] | 96 [88 to 99]
  Ser. Y - month 6 (n=24,24,24,25,23,72) | 96 [79 to 100] | 100 [86 to 100] | 96 [79 to 100] | 92 [74 to 99] | 4 [0 to 22] | 85 [74 to 92]
  Ser. Y - month 7 (n=25,24,24,25,22,72) | 100 [86 to 100] | 96 [79 to 100] | 100 [86 to 100] | 100 [86 to 100] | 14 [3 to 35] | 85 [74 to 92]

2. Primary Outcome: Percentages of Subjects With hSBA ≥1:5 Against Serogroup B Test Strains at One Month After Third Vaccination With One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Description: Antibody response was measured as the percentage of subjects with human serum bactericidal assay (hSBA) titers ≥1:5 and associated 95% CI, directed against to Serogroup B Test Strains at 6 months following first vaccine during the parent study NCT01210885 and one month after third vaccination (Month 7)
Time Frame: At month 6 and month 7
Population: Analysis was done by MITT Month 7 Set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 73
Percentages of subjects
  H44/76 (fHbp) - month 6 (n=25,24,25,24,23,72) | 40 [21 to 61] | 46 [26 to 67] | 52 [31 to 72] | 29 [13 to 51] | 35 [16 to 57] | 3 [0 to 10]
  H44/76 (fHbp) - month 7 (n=25,24,24,24,25,22,73) | 92 [74 to 99] | 96 [79 to 100] | 96 [79 to 100] | 92 [74 to 99] | 91 [71 to 99] | 4 [1 to 12]
  5/99 (NadA) - month 6 (n=25,24,24,25,23,72) | 96 [80 to 100] | 100 [86 to 100] | 96 [79 to 100] | 100 [86 to 100] | 100 [85 to 100] | 15 [8 to 26]
  5/99 (NadA) - month 7 (n=25,24,24,25,23,73) | 100 [86 to 100] | 100 [86 to 100] | 100 [86 to 100] | 100 [86 to 100] | 100 [85 to 100] | 16 [9 to 27]
  NZ98/254(PorA) - month 6 (n=25,24,24,25,23,72) | 12 [3 to 31] | 8 [1 to 27] | 29 [13 to 51] | 12 [3 to 31] | 9 [1 to 28] | 0 [0 to 5]
  NZ98/254(PorA) - month 7 (n=25,24,24,25,23,73) | 20 [7 to 41] | 29 [13 to 51] | 88 [68 to 97] | 76 [55 to 91] | 17 [5 to 39] | 1 [0.035 to 7]
  M14459(fHBP) - month 6 (n=25,24,25,25,23,71) | 24 [9 to 45] | 25 [10 to 47] | 32 [15 to 54] | 16 [5 to 36] | 17 [5 to 39] | 6 [2 to 14]
  M14459(fHBP) - month 7 (n=25,24,23,25,22,73) | 80 [59 to 93] | 79 [58 to 93] | 87 [66 to 97] | 88 [69 to 97] | 64 [41 to 83] | 8 [3 to 17]
  M07-0241084(NHBA) - month 6 (n=25,23,23,25,23,70) | 20 [7 to 41] | 35 [16 to 57] | 39 [20 to 61] | 52 [31 to 72] | 30 [13 to 53] | 30 [20 to 42]
  M07-0241084(NHBA) - month 7 (n=25,23,22,25,21,72) | 68 [46 to 85] | 61 [39 to 80] | 95 [77 to 100] | 92 [74 to 99] | 62 [38 to 82] | 29 [19 to 41]
  M01-0240364(NadA) - month 6 (n=25,21,24,24,21,71) | 16 [5 to 36] | 38 [18 to 62] | 25 [10 to 47] | 33 [16 to 55] | 33 [15 to 57] | 4 [1 to 12]
  M01-0240364(NadA) - month 7 (n=24,23,24,25,23,71) | 96 [79 to 100] | 100 [85 to 100] | 100 [86 to 100] | 96 [80 to 100] | 96 [78 to 100] | 4 [1 to 12]

3. Secondary Outcome: Geometric Mean Titers (GMT) for N Meningitidis Serogroups A, C, W and Y at One Month After the Third Vaccination With One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean hSBA Titers against N meningitidis Serogroups A, C, W and Y at One of Four MenABCWY Formulations or rMenB at 6 months following first vaccine during the parent study NCT01210885 and one month after third vaccination (Month 7)
Time Frame: At month 6 and month 7
Population: Analysis was done by MITT Month 7 Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 72
Titers
  Ser. A - month 6 (n=23,24,24,25,23,69) | 15 [6.66 to 33] | 44 [20 to 96] | 31 [14 to 68] | 21 [9.53 to 44] | 4.52 [2.02 to 10] | 21 [13 to 34]
  Ser. A - month 7 (n=24,24,21,25,22,71) | 247 [120 to 509] | 322 [157 to 659] | 242 [113 to 521] | 274 [136 to 553] | 135 [64 to 287] | 22 [14 to 33]
  Ser. C - month 6 (n=22,24,24,24,21,70) | 211 [125 to 355] | 153 [93 to 251] | 168 [102 to 278] | 137 [83 to 224] | 4.54 [2.66 to 7.75] | 25 [18 to 34]
  Ser. C - month 7 (n=23,24,23,25,22,72) | 796 [472 to 1343] | 716 [430 to 1193] | 670 [397 to 1130] | 634 [385 to 1044] | 31 [18 to 53] | 19 [14 to 26]
  Ser. W - month 6 (n=24,24,25,24,22,69) | 189 [116 to 305] | 184 [144 to 296] | 202 [127 to 324] | 164 [102 to 263] | 11 [6.67 to 18] | 128 [95 to 173]
  Ser. W - month 7 (n=23,24,21,25,21,72) | 710 [442 to 1143] | 695 [441 to 1096] | 929 [570 to 1512] | 684 [438 to 1069] | 126 [77 to 207] | 130 [98 to 172]
  Ser. Y - month 6 (n=24,24,24,25,23,72) | 203 [111 to 372] | 233 [128 to 425] | 158 [86 to 289] | 129 [72 to 233] | 1.72 [0.93 to 3.18] | 97 [67 to 140]
  Ser. Y - month 7 (n=25,24,24,25,22,72) | 695 [385 to 1255] | 629 [346 to 1144] | 619 [339 to 1129] | 432 [241 to 776] | 2.64 [1.41 to 4.96] | 85 [59 to 122]

4. Secondary Outcome: Geometric Mean Ratio (GMR) for (95%CI) for N Meningitidis Serogroups A, C, W and Y at One Month After the Third Vaccination With One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean Ratio (95% CI), against N meningitidis Serogroups A, C, W and Y at One Month After the Third Vaccination (month 7) With One of Four MenABCWY Formulations or rMenB
Time Frame: At month 7
Population: Analysis was done by MITT Month 7 Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 72
Ratio
  Ser. A (n=22,24,21,25,22,68) | 15 [8.88 to 25] | 7.53 [4.58 to 12] | 10 [6.1 to 18] | 14 [8.37 to 22] | 34 [20 to 57] | 1.05 [0.77 to 1.43]
  Ser. C (n=21,24,22,24,20,70) | 3.43 [2.59 to 4.54] | 4.63 [3.56 to 6.02] | 3.85 [2.92 to 5.06] | 5.01 [3.85 to 6.5] | 8.41 [6.31 to 11] | 0.75 [0.64 to 0.89]
  Ser. W (n=23,24,21,24,20,69) | 3.42 [2.41 to 4.85] | 3.66 [2.62 to 5.12] | 3.98 [2.78 to 5.69] | 4.05 [2.9 to 5.66] | 11 [7.55 to 16] | 1.01 [0.82 to 1.24]
  Ser. Y (n=24,24,23,25,22,71) | 3.33 [2.31 to 4.79] | 2.68 [1.87 to 3.85] | 4.45 [3.06 to 6.45] | 3.32 [2.33 to 4.73] | 1.46 [1 to 2.14] | 0.81 [0.65 to 1.02]

5. Secondary Outcome: GMT for N Meningitidis Against Serogroup B Test Strains at One Month After the Third Vaccination With One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean hSBA Titers Against Serogroup B Test Strains at 6 months following first vaccine during the parent study NCT01210885 and one month after third vaccination (Month 7) with One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Time Frame: At month 6 and month 7
Population: Analysis was done by MITT Month 7 Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 73
Titers
  H44/76 (fHbp) - month 6 (n=25,24,25,24,23,72) | 5.9 [3.07 to 11] | 6.88 [3.56 to 13] | 12 [6.14 to 23] | 5.25 [2.71 to 10] | 6.42 [3.27 to 13] | 1.18 [1.01 to 1.37]
  H44/76 (fHbp) - month 7 (n= 25,24,24,25,22,73) | 109 [60 to 201] | 154 [83 to 285] | 181 [97 to 336] | 114 [62 to 208] | 109 [57 to 209] | 1.21 [1.04 to 1.4]
  5/99 (NadA) - month 6 (n=25,24,24,25,23,72) | 78 [52 to 118] | 122 [80 to 186] | 46 [30 to 71] | 84 [56 to 127] | 152 [99 to 234] | 1.74 [1.36 to 2.22]
  5/99 (NadA) - month 7 (n=25,24,24,25,23,73) | 546 [365 to 817] | 740 [492 to 1112] | 665 [441 to 1002] | 527 [354 to 786] | 832 [548 to 1263] | 1.93 [1.5 to 2.48]
  NZ98/254(PorA) - month 6 (n=25,24,24,25,23,72) | 1.96 [1.29 to 3] | 1.85 [1.21 to 2.85] | 3.47 [2.26 to 5.35] | 1.89 [1.24 to 2.88] | 1.81 [1.17 to 2.81] | 1.15 [1.05 to 1.25]
  NZ98/254(PorA) - month 7 (n=25,24,24,25,23,72) | 2.37 [1.5 to 3.74] | 3.26 [2.06 to 5.17] | 24 [15 to 37] | 12 [7.57 to 19] | 2.64 [1.65 to 4.23] | 1.2 [1.07 to 1.33]
  M14459(fHBP) - month 6 (n=25,24,25,25,23,71) | 2.71 [1.72 to 4.27] | 3.29 [2.08 to 5.21] | 4.49 [2.85 to 7.06] | 2.34 [1.49 to 3.67] | 2.48 [1.55 to 3.97] | 1.28 [1.11 to 1.49]
  M14459(fHBP) - month 7 (n=25,24,23,25,22,73) | 16 [10 to 27] | 27 [17 to 44] | 45 [27 to 75] | 20 [13 to 33] | 12 [7.07 to 20] | 1.28 [1.1 to 1.49]
  M07-0241084(NHBA) - month 6 (n=25,23,23,25,23,70) | 3.37 [1.98 to 5.73] | 3.66 [2.12 to 6.34] | 6.92 [3.99 to 12] | 6.45 [3.81 to 11] | 3.32 [1.91 to 5.75] | 2.99 [2.16 to 4.14]
  M07-0241084(NHBA) - month 7 (n=25,23,22,25,21,72) | 12 [7.07 to 21] | 9.48 [5.37 to 17] | 38 [21 to 69] | 25 [15 to 44] | 9.73 [5.33 to 18] | 3.03 [2.22 to 4.15]
  M01-0240364 (NadA) - month 6 (n=25,21,23,24,21,71) | 4.62 [2.15 to 9.95] | 9.98 [4.37 to 23] | 6.95 [3.19 to 15] | 7.44 [3.44 to 16] | 7.21 [3.15 to 17] | 1.18 [1 to 1.39]
  M01-0240364 (NadA) - month 7 (n=24,23,23,25,23,71) | 311 [152 to 637] | 533 [259 to 1098] | 385 [188 to 786] | 286 [143 to 573] | 474 [229 to 980] | 1.18 [1 to 1.39]

6. Secondary Outcome: GMR for (95%CI) for N Meningitidis Against Serogroup B Test Strains at One Month After the Third Vaccination With One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean Ratio (95% CI), against Serogroup B Test Strains at One Month After the Third Vaccination (month 7) with One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Time Frame: At month 7
Population: Analysis was done by MITT Month 7 Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 73
Ratio
  H44/76 (fHbp) (n=25,24,24,24,22,72) | 18 [12 to 29] | 22 [14 to 36] | 14 [8.88 to 23] | 22 [14 to 36] | 16 [9.83 to 26] | 1.03 [0.98 to 1.08]
  5/99 (NadA) (n=25,24,23,25,23,72) | 6.96 [5.15 to 9.42] | 6.04 [4.45 to 8.21] | 14 [11 to 20] | 6.25 [4.63 to 8.44] | 5.47 [4 to 7.48] | 1.12 [0.93 to 1.36]
  NZ98/254 (PorA) (n=25,24,23,25,23,72) | 1.21 [0.87 to 1.67] | 1.76 [1.26 to 2.45] | 6.56 [4.67 to 9.2] | 6.29 [4.55 to 8.69] | 1.45 [1.04 to 2.04] | 1.05 [0.95 to 1.15]
  M14459 (fHBP) (n=25,24,23,25,22,71) | 5.99 [4.11 to 8.73] | 8.1 [5.54 to 12] | 9.08 [6.14 to 13] | 8.58 [5.91 to 12] | 4.37 [2.93 to 6.53] | 1.01 [0.91 to 1.11]
  M07-0241084 (NHBA) (n=25,22,20,25,21,69) | 3.61 [2.57 to 5.09] | 2.46 [1.71 to 3.54] | 5.18 [3.53 to 7.58] | 3.92 [2.8 to 5.51] | 2.75 [1.89 to 4.01] | 1.01 [0.91 to 1.12]
  M01-0240364 (NadA) (n=24,20,23,24,21,69) | 65 [37 to 114] | 50 [27 to 92] | 65 [37 to 116] | 40 [23 to 71] | 66 [36 to 120] | 1 [0.97 to 1.04]

7. Secondary Outcome: Percentages of Subjects With Seroresponse Against N Meningitidis Serogroups A, C, W and Y at 1 Month After the Third Vaccination With One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Description: Antibody response was measured as the percentage of subjects with seroresponse Against N meningitidis Serogroups A, C, W and Y, after pre and post vaccination at month 6 and after the third vaccination (month 7) with One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo. Seroresponse to N meningitidis serogroups A, C, W and Y is defined as: For subjects with a prevaccination hSBA <1:4, a postvaccination hSBA ≥1:8;For subjects with a prevaccination hSBA ≥1:4, an increase in hSBA titer of at least four times the prevaccination titer.
Time Frame: At month 7
Population: Analysis was done by MITT month 7 Set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 71
Percentages of subjects
  Ser. A (n=22,24,21,25,22,68) | 59 [36 to 79] | 67 [45 to 84] | 67 [43 to 85] | 72 [51 to 88] | 82 [60 to 95] | 3 [0 to 10]
  Ser. C (n=21,24,22,24,20,70) | 48 [26 to 70] | 54 [33 to 74] | 59 [36 to 79] | 67 [45 to 84] | 60 [36 to 81] | 0 [0 to 5]
  Ser. W (n=23,24,21,24,20,69) | 35 [16 to 57] | 38 [19 to 59] | 48 [26 to 70] | 58 [37 to 78] | 60 [36 to 81] | 3 [0 to 10]
  Ser. Y (n=24,24,23,25,22,71) | 29 [13 to 51] | 38 [19 to 59] | 43 [23 to 66] | 32 [15 to 54] | 5 [0 to 23] | 0 [0 to 5]

8. Secondary Outcome: Percentages of Subjects With 4-fold Increase in hSBA Titers Against Serogroup B Test Strains at One Month After Third Vaccination With One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Description: Antibody response was measured as the percentage of subjects with 4-fold Increase in human serum bactericidal assay (hSBA) titers and associated 95% CI, Against Serogroup B Test Strains at One Month After Third Vaccination (month 7) with One of Four MenABCWY Formulations, rMenB or MenACWY/Placebo
Time Frame: At month 7
Population: Analysis was done by MITT month 7 Set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 24 | 25 | 23 | 72
Percentages of subjects
  H44/76 (fHbp) (n=25,24,24,24,22,72) | 80 [59 to 93] | 88 [68 to 97] | 83 [63 to 95] | 88 [68 to 97] | 73 [50 to 89] | 0 [0 to 5]
  5/99 (NadA) (n=25,24,23,25,23,72) | 80 [59 to 93] | 67 [45 to 84] | 83 [61 to 95] | 76 [55 to 91] | 57 [34 to 77] | 3 [0 to 10]
  NZ98/254 (PorA) (n=25,24,23,25,23,72) | 4 [0 to 20] | 17 [5 to 37] | 61 [39 to 80] | 44 [24 to 65] | 17 [5 to 39] | 1 [0.035 to 7]
  M14459 (fHBP) (n=25,24,23,25,22,71) | 56 [35 to 76] | 54 [33 to 74] | 65 [43 to 84] | 52 [31 to 72] | 50 [28 to 72] | 1 [0.036 to 8]
  M07-0241084 (NHBA) (n=25,22,20,25,21,69) | 36 [18 to 57] | 23 [8 to 45] | 60 [36 to 81] | 44 [24 to 65] | 29 [11 to 52] | 0 [0 to 5]
  M01-0240364 (NadA) (n=24,20,23,24,21,69) | 88 [68 to 97] | 80 [56 to 94] | 83 [61 to 95] | 79 [58 to 93] | 90 [70 to 99] | 0 [0 to 5]

9. Secondary Outcome: GMT for N Meningitidis Serogroups A, C, W and Y at Month 0 Through Month 12 Following Vaccination at Month 0, Month 2 With One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean hSBA Titers Against N meningitidis Serogroups A, C, W and Y after first (month 1) and second (month 3) vaccination during the parent study NCT01210885, after 6 month of the first vaccination (6 month) in the parent study and after the third vaccination (month 7) and 6 month after the third vaccination (month 12) with One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo.
Time Frame: At month 1, 3, 6, 7 and 12
Population: Analysis was done by MITT Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 2 B: Two doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine in previous study and one dose of Tdap in current study
Arm/Group | 2ABCWY | 2ABx2CWY | 2ABCWY+OMV | 2ABCWYqOMV | 2 B | 1ACWY
Number analyzed (Participants) | 49 | 48 | 48 | 49 | 50 | 73
Titers
  Ser. A - month 1 (n=48,48,47,49,50,70) | 61 [35 to 107] | 61 [35 to 107] | 49 [28 to 86] | 37 [21 to 65] | 2.96 [1.71 to 5.13] | 107 [66 to 172]
  Ser. A - month 3 (n=49,48,47,48,50,72) | 162 [106 to 249] | 206 [134 to 316] | 183 [118 to 282] | 169 [109 to 262] | 44 [29 to 68] | 36 [25 to 52]
  Ser. A - month 6 (n=46,46,48,44,49,69) | 28 [16 to 49] | 44 [25 to 78] | 21 [12 to 36] | 24 [14 to 44] | 4.22 [2.43 to 7.33] | 20 [12 to 32]
  Ser. A - month 7 (n=48,47,46,49,50,71) | 24 [14 to 39] | 28 [17 to 46] | 17 [9.94 to 28] | 17 [10 to 29] | 3.18 [1.95 to 5.19] | 21 [13 to 31]
  Ser. A - month 12 (n=43,44,45,46,50,71) | 10 [5.69 to 18] | 9.73 [5.6 to 17] | 8.88 [5.09 to 15] | 8.08 [4.64 to 14] | 2.21 [1.31 to 3.75] | 14 [9.03 to 22]
  Ser. C - month 1 (n=48,48,48,48,50,71) | 51 [33 to 80] | 116 [75 to 180] | 99 [64 to 155] | 101 [64 to 159] | 8.76 [5.63 to 14] | 75 [51 to 109]
  Ser. C - month 3 (n=49,47,46,48,50,71) | 340 [252 to 460] | 501 [370 to 680] | 338 [248 to 461] | 380 [278 to 520] | 17 [12 to 22] | 45 [35 to 58]
  Ser. C - month 6 (n=46,48,47,48,49,70) | 133 [94 to 189] | 186 [133 to 261] | 117 [83 to 165] | 157 [111 to 223] | 6.77 [4.82 to 9.52] | 23 [17 to 31]
  Ser. C - month 7 (n=48,47,46,49,50,72) | 110 [78 to 156] | 153 [108 to 217] | 88 [61 to 126] | 128 [90 to 183] | 5.53 [3.9 to 7.84] | 18 [13 to 24]
  Ser. C - month 12 (n=44,46,46,46,50,72) | 55 [38 to 81] | 66 [45 to 95] | 45 [31 to 65] | 72 [49 to 105] | 6.03 [4.19 to 8.69] | 14 [10 to 19]
  Ser. W - month 1 (n=48,48,47,48,49,72) | 163 [113 to 237] | 243 [168 to 352] | 173 [119 to 252] | 233 [160 to 341] | 29 [20 to 42] | 210 [154 to 287]
  Ser. W - month 3 (n=49,46,47,48,50,72) | 370 [290 to 472] | 514 [400 to 661] | 349 [272 to 448] | 435 [338 to 559] | 140 [110 to 179] | 166 [135 to 204]
  Ser. W - month 6 (n=44,47,45,45,43,69) | 202 [144 to 284] | 196 [141 to 272] | 143 [102 to 200] | 194 [138 to 274] | 15 [11 to 21] | 117 [88 to 154]
  Ser. W - month 7 (n=46,47,45,47,45,72) | 173 [125 to 240] | 167 [121 to 230] | 118 [85 to 164] | 168 [121 to 234] | 13 [9.72 to 19] | 121 [93 to 159]
  Ser. W - month 12 (n=45,45,45,43,46,69) | 119 [82 to 174] | 113 [77 to 164] | 83 [57 to 120] | 109 [73 to 161] | 11 [7.81 to 17] | 75 [55 to 103]
  Ser. Y - month 1 (n=48,48,48,49,49,73) | 98 [66 to 145] | 119 [80 to 177] | 76 [51 to 113] | 92 [62 to 136] | 5.6 [3.77 to 8.32] | 92 [66 to 128]
  Ser. Y - month 3 (n=49,48,47,49,50,73) | 214 [162 to 281] | 283 [215 to 374] | 195 [147 to 258] | 226 [172 to 298] | 4.7 [3.58 to 6.18] | 72 [57 to 91]
  Ser. Y - month 6 (n=48,48,48,48,49,72) | 206 [134 to 315] | 249 [162 to 382] | 138 [90 to 212] | 154 [100 to 237] | 1.93 [1.26 to 2.95] | 84 [58 to 120]
  Ser. Y - month 7 (n=46,48,46,49,50,72) | 180 [116 to 278] | 213 [139 to 327] | 100 [65 to 155] | 127 [83 to 194] | 2.05 [1.34 to 3.13] | 75 [52 to 108]
  Ser. Y - month 12 (n=45,47,45,46,50,70) | 88 [55 to 141] | 112 [71 to 178] | 55 [34 to 88] | 75 [47 to 121] | 1.59 [1.01 to 2.5] | 47 [31 to 69]

10. Secondary Outcome: GMR for N Meningitidis Serogroups A, C, W and Y at Month 0 Through Month 12 Following Vaccination at Month 0, Month 2 With One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean Ratios (95%CI) Against N meningitidis Serogroups A, C, W and Y after after first (month 1) and second (month 3) vaccination during the parent study NCT01210885, after 6 month of the first vaccination (6 month) in the parent study and after the third vaccination (month 7) and 6 month after the third vaccination (month 12) with One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Time Frame: At month 1, 3, 6, 7 and 12
Population: Analysis was done by Per MITT Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 2ABCWY | 2ABx2CWY | 2ABCWY+OMV | 2ABCWYqOMV | 2 B | 1ACWY
Number analyzed (Participants) | 49 | 48 | 48 | 49 | 50 | 73
Ratio
  Ser. A - month 1 (n=48,48,47,48,50,70) | 41 [23 to 73] | 45 [26 to 80] | 36 [20 to 65] | 30 [17 to 53] | 2.25 [1.28 to 3.93] | 78 [48 to 127]
  Ser. A - month 3 (n=49,48,47,47,50,72) | 107 [68 to 168] | 150 [95 to 235] | 135 [85 to 214] | 137 [86 to 217] | 34 [21 to 52] | 26 [18 to 38]
  Ser. A - month 6 (n=46,46,48,44,49,69) | 19 [11 to 34] | 32 [18 to 57] | 15 [8.77 to 27] | 20 [11 to 35] | 3.19 [1.85 to 5.59] | 15 [9.12 to 24]
  Ser. A - month 7 (n=48,47,46,48,50,71) | 16 [9.83 to 27] | 21 [12 to 34] | 12 [7.36 to 21] | 14 [8.22 to 23] | 2.41 [1.47 to 3.97] | 15 [9.87 to 23]
  Ser. A - month 12 (n=43,44,45,45,50,71) | 6.97 [3.93 to 12] | 7.18 [4.11 to 13] | 6.61 [3.77 to 12] | 6.42 [3.67 to 11] | 1.68 [0.99 to 2.85] | 11 [6.65 to 17]
  Ser. C - month 1 (n=48,48,48,47,50,70) | 11 [6.83 to 19] | 26 [16 to 43] | 19 [12 to 31] | 20 [12 to 33] | 1.42 [0.87 to 2.32] | 16 [11 to 25]
  Ser. C - month 3 (n=49,47,46,46,50,70) | 72 [47 to 110] | 114 [74 to 175] | 60 [39 to 93] | 71 [45 to 110] | 2.36 [1.54 to 3.59] | 9.54 [6.61 to 14]
  Ser. C - month 6 (n=46,48,47,46,49,69) | 29 [19 to 45] | 41 [27 to 63] | 22 [14 to 34] | 31 [20 to 47] | 1.07 [0.7 to 1.63] | 5.14 [3.57 to 7.39]
  Ser. C - month 7 (n=48,47,46,47,50,71) | 24 [16 to 37] | 33 [21 to 51] | 16 [10 to 25] | 25 [16 to 38] | 0.85 [0.55 to 1.3] | 3.9 [2.7 to 5.64]
  Ser. C - month 12 (n=44,46,46,44,50,71) | 12 [7.82 to 19] | 16 [10 to 24] | 8.88 [5.7 to 14] | 15 [9.57 to 24] | 0.99 [0.65 to 1.52] | 3.06 [2.12 to 4.4]
  Ser. W - month 1 (n=48,47,47,46,49,72) | 9.2 [5.41 to 16] | 13 [7.42 to 21] | 7.41 [4.34 to 13] | 10 [6.1 to 18] | 1.15 [0.68 to 1.95] | 10 [6.49 to 16]
  Ser. W - month 3 (n=49,45,47,46,50,72) | 20 [11 to 34] | 27 [15 to 48] | 12 [6.7 to 21] | 19 [11 to 35] | 4.83 [2.76 to 8.46] | 7.32 [4.53 to 12]
  Ser. W - month 6 (n=44,46,45,43,43,69) | 11 [6.33 to 20] | 9.75 [5.64 to 17] | 5.44 [3.11 to 9.52] | 9.75 [5.51 to 17] | 0.58 [0.33 to 1.02] | 5.17 [3.25 to 8.24]
  Ser. W - month 7 (n=46,46,45,45,45,72) | 9.21 [5.2 to 16] | 8.17 [4.64 to 14] | 4.84 [2.72 to 8.62] | 7.94 [4.44 to 14] | 0.55 [0.31 to 0.97] | 5.47 [3.4 to 8.8]
  Ser. W - month 12 (n=45,44,45,42,46,69) | 7.33 [4.08 to 13] | 6.54 [3.62 to 12] | 3.52 [1.95 to 6.33] | 4.83 [2.62 to 8.92] | 0.49 [0.27 to 0.89] | 3.62 [2.21 to 5.94]
  Ser. Y - month 1 (n=48,47,48,49,49,73) | 21 [13 to 32] | 26 [17 to 40] | 15 [9.89 to 24] | 20 [13 to 31] | 1.02 [0.66 to 1.58] | 16 [11 to 23]
  Ser. Y - month 3 (n=49,47,47,49,50,73) | 44 [30 to 63] | 59 [41 to 85] | 37 [25 to 54] | 47 [33 to 68] | 0.8 [0.56 to 1.15] | 12 [8.54 to 16]
  Ser. Y - month 6 (n=48,47,48,48,49,72) | 44 [27 to 71] | 56 [34 to 91] | 27 [16 to 44] | 33 [20 to 54] | 0.35 [0.21 to 0.56] | 14 [9.04 to 21]
  Ser. Y - month 7 (n=46,47,46,49,50,72) | 37 [22 to 61] | 45 [27 to 74] | 19 [11 to 31] | 26 [16 to 43] | 0.35 [0.21 to 0.56] | 12 [7.76 to 18]
  Ser. Y - month 12 (n=45,46,45,46,50,70) | 18 [11 to 31] | 25 [15 to 42] | 10 [6.14 to 18] | 16 [9.64 to 28] | 0.27 [0.16 to 0.45] | 7.27 [4.68 to 11]

11. Secondary Outcome: GMT Against Serogroup B Test Strains at Month 0 Through Month 12 Following Vaccination at Month 0 and Month 2 With One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean hSBA Titers Against Serogroup B Test Strains after first (month 1) and second (month 3) vaccination during the parent study NCT01210885, After Third Vaccination (month 7) and 6 month after the third vaccination (month 12) with One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Time Frame: At month 1, 3, 6, 7 and 12
Population: Analysis was done by MITT Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 2ABCWY | 2ABx2CWY | 2ABCWY+OMV | 2ABCWYqOMV | 2 B | 1ACWY
Number analyzed (Participants) | 49 | 49 | 48 | 49 | 50 | 73
Titers
  H44/76 (fHbp) - month 1 (n=48,48,48,49,50,73) | 5.56 [3.44 to 8.99] | 10 [6.38 to 17] | 15 [9.5 to 25] | 11 [6.93 to 18] | 4.56 [2.84 to 7.3] | 1.51 [1.19 to 1.92]
  H44/76 (fHbp) - month 3 (n=49,48,46,48,50,72) | 74 [53 to 102] | 114 [82 to 158] | 114 [81 to 159] | 133 [96 to 186] | 44 [32 to 61] | 1.27 [1.07 to 1.5]
  H44/76 (fHbp) - month 6 (n=47,48,48,48,50,72) | 7.87 [5.04 to 12] | 7.76 [4.98 to 12] | 9.44 [6.04 to 15] | 14 [9.2 to 23] | 4.34 [2.81 to 6.71] | 1.18 [1.01 to 1.37]
  H44/76 (fHbp) - month 7 (n=48,48,47,49,49,73) | 4.62 [3.04 to 7.02] | 5.75 [3.79 to 8.73] | 6.12 [4 to 9.37] | 11 [7.15 to 17] | 3.55 [2.35 to 5.37] | 1.21 [1.04 to 1.4]
  H44/76 (fHbp) - month 12 (n=45,47,45,46,50,71) | 3.24 [2.18 to 4.8] | 2.31 [1.57 to 3.39] | 4 [2.69 to 5.97] | 4.31 [2.91 to 6.4] | 2.42 [1.66 to 3.52] | 1.13 [1 to 1.29]
  5/99 (NadA) - month 1 (n=48,48,47,49,50,72) | 44 [29 to 65] | 91 [62 to 135] | 23 [15 to 34] | 34 [23 to 51] | 58 [39 to 85] | 2.27 [1.82 to 2.85]
  5/99 (NadA) - month 3 (n=49,48,47,47,50,71) | 257 [203 to 324] | 401 [318 to 507] | 337 [266 to 427] | 363 [285 to 462] | 322 [255 to 406] | 2.11 [1.65 to 2.7]
  5/99 (NadA) - month 6 (n=47,49,48,48,48,72) | 69 [51 to 93] | 122 [91 to 163] | 55 [41 to 74] | 72 [53 to 97] | 73 [54 to 98] | 1.74 [1.36 to 2.22]
  5/99 (NadA) - month 7 (n=47,48,47,49,50,73) | 55 [42 to 73] | 96 [72 to 127] | 44 [33 to 58] | 59 [45 to 79] | 68 [51 to 90] | 1.93 [1.5 to 2.48]
  5/99 (NadA) - month 12 (n=45,47,46,46,50,72) | 31 [22 to 44] | 46 [33 to 64] | 30 [21 to 42] | 35 [25 to 49] | 32 [23 to 44] | 1.53 [1.25 to 1.88]
  NZ98/254 (PorA) - month 1 (n=48,48,48,49,50,72) | 2.14 [1.58 to 2.9] | 2.42 [1.8 to 3.26] | 4.95 [3.66 to 6.7] | 4.26 [3.15 to 5.77] | 2.01 [1.49 to 2.71] | 1.51 [1.32 to 1.74]
  NZ98/254 (PorA) - month 3 (n=49,48,47,48,50,72) | 2.98 [2.18 to 4.06] | 3.86 [2.83 to 5.26] | 14 [10 to 19] | 12 [8.96 to 17] | 2.81 [2.06 to 3.84] | 1.49 [1.29 to 1.72]
  NZ98/254 (PorA) - month 6 (n=48,49,48,48,49,72) | 1.7 [1.28 to 2.26] | 1.88 [1.42 to 2.48] | 3.19 [2.4 to 4.25] | 3.09 [2.31 to 4.13] | 1.47 [1.1 to 1.95] | 1.15 [1.05 to 1.25]
  NZ98/254 (PorA) - month 7 (n=47,48,47,49,50,73) | 1.45 [1.05 to 2] | 1.76 [1.29 to 2.41] | 2.62 [1.9 to 3.62] | 2.49 [1.81 to 3.43] | 1.45 [1.06 to 2] | 1.2 [1.07 to 1.33]
  NZ98/254 (PorA) - month 12 (n=45,47,46,46,50,72) | 1.57 [1.2 to 2.06] | 1.6 [1.23 to 2.09] | 2.47 [1.89 to 3.24] | 2.18 [1.66 to 2.86] | 1.21 [0.93 to 1.57] | 1.15 [1.05 to 1.25]
  M14459 (fHBP) - month 1 (n=48,48,47,49,50,72) | 1.99 [1.44 to 2.75] | 2.66 [1.92 to 3.68] | 4.59 [3.28 to 6.44] | 3.47 [2.47 to 4.89] | 2.02 [1.46 to 2.8] | 1.26 [1.08 to 1.47]
  M14459 (fHBP) - month 3 (n=49,48,45,43,50,70) | 6.31 [4.28 to 9.32] | 13 [8.91 to 20] | 17 [11 to 26] | 20 [13 to 30] | 5.04 [3.39 to 7.47] | 1.29 [1.1 to 1.51]
  M14459 (fHBP) - month 6 (n=47,47,48,48,50,71) | 2.1 [1.59 to 2.79] | 2.63 [1.99 to 3.49] | 3.33 [2.49 to 4.44] | 3.15 [2.35 to 4.24] | 2.05 [1.55 to 2.71] | 1.28 [1.11 to 1.49]
  M14459 (fHBP) - month 7 (n=47,48,47,49,50,73) | 1.79 [1.29 to 2.49] | 2.4 [1.74 to 3.33] | 2.75 [1.96 to 3.86] | 3.59 [2.55 to 5.06] | 1.87 [1.35 to 2.59] | 1.28 [1.1 to 1.49]
  M14459 (fHBP) - month 12 ( n=45,47,45,47,50,72) | 1.73 [1.31 to 2.27] | 1.64 [1.25 to 2.14] | 2.43 [1.83 to 3.23] | 2.53 [1.91 to 3.36] | 1.44 [1.1 to 1.87] | 1.37 [1.15 to 1.64]
  M07-0241084 (NHBA) - month 1 (n=48,48,48,48,50,72) | 2.88 [2.17 to 3.81] | 3.17 [2.39 to 4.21] | 7.11 [5.18 to 9.76] | 5.51 [4.12 to 7.36] | 3.76 [2.85 to 4.97] | 2.68 [1.93 to 3.7]
  M07-0241084 (NHBA) - month 3 (n=48,48,42,45,49,68) | 4.34 [3.27 to 5.75] | 6.27 [4.71 to 8.33] | 12 [8.71 to 17] | 14 [10 to 19] | 6.25 [4.71 to 8.28] | 2.85 [2.08 to 3.91]
  M07-0241084 (NHBA) - month 6 (n=47,48,48,48,49,70) | 3.78 [2.88 to 4.95] | 3.3 [2.51 to 4.34] | 5.43 [4 to 7.37] | 6.93 [5.23 to 9.19] | 3.36 [2.56 to 4.4] | 2.99 [2.16 to 4.14]
  M07-0241084 (NHBA) - month 7 (n=47,48,47,48,50,72) | 3.51 [2.54 to 4.85] | 3.19 [2.3 to 4.41] | 5.18 [3.58 to 7.48] | 6.58 [4.7 to 9.22] | 3.78 [2.74 to 5.2] | 3.03 [2.22 to 4.15]
  M07-0241084(NHBA) - month 12 (n=45,46,45,47,50,70) | 3.71 [2.74 to 5.03] | 2.82 [2.08 to 3.83] | 4.92 [3.51 to 6.89] | 6.16 [4.53 to 8.38] | 3.09 [2.31 to 4.14] | 2.91 [2.06 to 4.12]
  M01-0240364 (NadA) - month 1 (n=48,44,46,48,50,72) | 5.46 [3.1 to 9.61] | 6.42 [3.54 to 12] | 4.7 [2.58 to 8.58] | 4.24 [2.33 to 7.71] | 4.25 [2.44 to 7.41] | 1.12 [0.98 to 1.29]
  M01-0240364 (NadA) - month 3 (n=48,48,44,42,49,70) | 67 [38 to 118] | 192 [109 to 339] | 133 [72 to 245] | 125 [67 to 233] | 88 [50 to 154] | 1.41 [1.07 to 1.85]
  M01-0240364 (NadA) - month 6 (n=46,48,48,48,48,71) | 8.59 [4.95 to 15] | 17 [9.65 to 29] | 11 [6.48 to 20] | 6.27 [3.52 to 11] | 7.02 [4.07 to 12] | 1.18 [1 to 1.39]
  M01-0240364 (NadA) - month 7 (n=44,48,48,48,50,71) | 5.38 [3.2 to 9.03] | 9.65 [5.83 to 16] | 7.51 [4.45 to 13] | 4.13 [2.43 to 7.01] | 5.72 [3.49 to 9.35] | 1.18 [1 to 1.39]
  M01-0240364 (NadA) - month12 (n=43,45,44,44,50,72) | 3.85 [2.16 to 6.84] | 4.79 [2.72 to 8.44] | 5.76 [3.19 to 10] | 3.23 [1.78 to 5.87] | 2.88 [1.68 to 4.92] | 1.15 [0.97 to 1.37]

12. Secondary Outcome: GMR Against Serogroup B Test Strains at Month 0 Through Month 12 Following Vaccination at Month 0 and Month 2 With One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean Ratios (95%CI) Against Serogroup B Test Strains after first (month 1) and second (month 3) vaccination during the parent study NCT01210885, after 6 month of the first vaccination (month 6) in the parent study and after the third vaccination (month 7) and 6 month after the third vaccination (month 12) with One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Time Frame: At month 1, 3, 6, 7 and 12
Population: Analysis was done by MITT Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 2ABCWY | 2ABx2CWY | 2ABCWY+OMV | 2ABCWYqOMV | 2 B | 1ACWY
Number analyzed (Participants) | 49 | 49 | 48 | 49 | 50 | 73
Ratio
  H44/76 (fHbp) - month 1 (n=48,47,47,48,50,73) | 4.42 [2.73 to 7.16] | 7.99 [4.95 to 13] | 12 [7.44 to 20] | 8.82 [5.43 to 14] | 3.53 [2.2 to 5.65] | 1.15 [0.98 to 1.35]
  H44/76 (fHbp) - month 3 (n=49,47,45,47,50,72) | 61 [42 to 87] | 84 [58 to 121] | 87 [60 to 127] | 103 [71 to 150] | 32 [22 to 46] | 1.05 [0.89 to 1.24]
  H44/76 (fHbp) - month 6 (n=47,47,47,47,50,72) | 6.3 [4.01 to 9.9] | 5.94 [3.79 to 9.3] | 7.37 [4.69 to 12] | 11 [7.14 to 18] | 3.31 [2.13 to 5.14] | 0.89 [0.78 to 1.02]
  H44/76 (fHbp) - month 7 (n=48,47,46,48,49,73) | 3.73 [2.43 to 5.75] | 4.34 [2.82 to 6.68] | 4.75 [3.06 to 7.37] | 8.48 [5.49 to 13] | 2.66 [1.73 to 4.08] | 0.92 [0.79 to 1.06]
  H44/76 (fHbp) - month 12 (n=45,46,44,45,50,71) | 2.58 [1.73 to 3.84] | 1.77 [1.2 to 2.61] | 3.11 [2.08 to 4.66] | 3.41 [2.29 to 5.09] | 1.85 [1.27 to 2.71] | 0.86 [0.73 to 1.01]
  5/99 (NadA) - month 1 (n=48,48,47,48,50,72) | 18 [12 to 29] | 42 [27 to 65] | 12 [7.41 to 18] | 16 [10 to 26] | 21 [13 to 33] | 1 [0.85 to 1.18]
  5/99 (NadA) - month 3 (n=49,48,47,46,50,71) | 106 [74 to 151] | 184 [129 to 263] | 176 [122 to 253] | 174 [120 to 252] | 107 [75 to 153] | 1 [0.8 to 1.26]
  5/99 (NadA) - month 6 (n=47,49,48,47,48,72) | 28 [19 to 41] | 56 [39 to 82] | 29 [20 to 42] | 35 [24 to 51] | 25 [17 to 37] | 0.78 [0.61 to 0.99]
  5/99 (NadA) - month 7 (n=47,48,47,48,50,73) | 23 [16 to 34] | 44 [30 to 63] | 23 [16 to 33] | 29 [20 to 42] | 23 [16 to 34] | 0.86 [0.68 to 1.08]
  5/99 (NadA) - month 12 (n=45,47,46,45,50,72) | 13 [8.78 to 20] | 21 [14 to 31] | 15 [10 to 23] | 18 [12 to 28] | 11 [7.48 to 16] | 0.7 [0.59 to 0.83]
  NZ98/254(PorA) - month 1 (n=48,48,48,48,50,72) | 1.27 [0.93 to 1.73] | 1.46 [1.07 to 1.98] | 2.91 [2.14 to 3.96] | 2.51 [1.84 to 3.42] | 1.08 [0.8 to 1.46] | 1 [0.87 to 1.16]
  NZ98/254(PorA) - month 3 (n=49,48,47,47,50,72) | 1.74 [1.26 to 2.4] | 2.33 [1.69 to 3.21] | 8.25 [5.95 to 11] | 7.17 [5.16 to 9.96] | 1.46 [1.06 to 2.01] | 0.99 [0.83 to 1.17]
  NZ98/254(PorA) - month 6 (n=48,49,48,47,49,72) | 0.99 [0.73 to 1.33] | 1.14 [0.85 to 1.53] | 1.86 [1.38 to 2.52] | 1.79 [1.32 to 2.44] | 0.75 [0.56 to 1.02] | 0.76 [0.65 to 0.89]
  NZ98/254(PorA) - month 7 (n=47,48,47,48,50,73) | 0.85 [0.61 to 1.19] | 1.07 [0.76 to 1.49] | 1.53 [1.09 to 2.15] | 1.45 [1.03 to 2.03] | 0.73 [0.52 to 1.01] | 0.8 [0.67 to 0.94]
  NZ98/254(PorA) - month 12 (n=45,47,46,45,50,72) | 0.91 [0.68 to 1.22] | 0.97 [0.73 to 1.29] | 1.41 [1.05 to 1.88] | 1.25 [0.93 to 1.68] | 0.6 [0.46 to 0.8] | 0.77 [0.66 to 0.9]
  M14459(fHBP) - month 1 (n=48,47,44,45,50,71) | 1.57 [1.13 to 2.17] | 2.09 [1.51 to 2.89] | 3.61 [2.58 to 5.06] | 2.73 [1.95 to 3.84] | 1.57 [1.14 to 2.16] | 0.95 [0.87 to 1.03]
  M14459(fHBP) - month 3 (n=49,47,42,41,50,69) | 4.96 [3.35 to 7.36] | 10 [6.77 to 15] | 13 [8.66 to 20] | 15 [9.83 to 23] | 3.54 [2.4 to 5.23] | 1.04 [0.9 to 1.2]
  M14459(fHBP) - month 6 (n=47,46,45,44,50,70) | 1.65 [1.25 to 2.19] | 2.04 [1.54 to 2.71] | 2.58 [1.94 to 3.45] | 2.46 [1.83 to 3.31] | 1.53 [1.16 to 2.02] | 0.99 [0.87 to 1.12]
  M14459(fHBP) - month 7 (n=47,47,44,45,50,72) | 1.4 [1 to 1.96] | 1.82 [1.31 to 2.54] | 2.08 [1.48 to 2.94] | 2.75 [1.95 to 3.9] | 1.3 [0.94 to 1.8] | 0.97 [0.83 to 1.13]
  M14459(fHBP) - month 12 (n=45,46,42,43,50,71) | 1.35 [1.02 to 1.77] | 1.26 [0.96 to 1.65] | 1.86 [1.4 to 2.47] | 1.96 [1.48 to 2.61] | 1.05 [0.81 to 1.37] | 1.03 [0.87 to 1.24]
  M07-0241084(NHBA) - month 1 (n=47,45,37,44,50,66) | 1.07 [0.81 to 1.42] | 1.14 [0.86 to 1.52] | 2.6 [1.89 to 3.57] | 2.03 [1.52 to 2.73] | 1.31 [1 to 1.72] | 1.02 [0.87 to 1.19]
  M07-0241084(NHBA) - month 3 (n=47,45,33,40,49,65) | 1.62 [1.19 to 2.19] | 2.1 [1.55 to 2.85] | 4.46 [3.11 to 6.39] | 4.94 [3.56 to 6.84] | 1.91 [1.42 to 2.56] | 1.13 [0.89 to 1.44]
  M07-0241084(NHBA) - month 6 (n=46,45,37,43,49,65) | 1.39 [1.04 to 1.85] | 1.13 [0.85 to 1.5] | 1.91 [1.39 to 2.64] | 2.53 [1.88 to 3.4] | 1.07 [0.81 to 1.42] | 1.2 [0.97 to 1.49]
  M07-0241084(NHBA) - month 7(n=46,45,36,43,50,66) | 1.29 [0.91 to 1.82] | 1.05 [0.74 to 1.48] | 1.81 [1.22 to 2.68] | 2.41 [1.68 to 3.46] | 1.12 [0.8 to 1.57] | 1.21 [0.96 to 1.51]
  M07-0241084(NHBA) - month 12 (n=44,43,36,43,50,64) | 1.38 [0.99 to 1.9] | 0.94 [0.68 to 1.3] | 1.7 [1.18 to 2.43] | 2.24 [1.61 to 3.12] | 0.94 [0.69 to 1.28] | 1.19 [0.9 to 1.58]
  M01-0240364(NadA) - month 1 (n=48,42,42,44,50,71) | 4.42 [2.51 to 7.77] | 5.08 [2.8 to 9.2] | 3.77 [2.07 to 6.88] | 3.35 [1.84 to 6.08] | 3.35 [1.93 to 5.83] | 1 [0.86 to 1.16]
  M01-0240364(NadA) - month 3 (n=48,46,40,40,49,69) | 57 [32 to 102] | 145 [80 to 261] | 105 [56 to 199] | 89 [47 to 170] | 64 [36 to 113] | 1.28 [1.01 to 1.63]
  M01-0240364(NadA) - month 6 (n=46,46,44,44,48,70) | 7.07 [4.05 to 12] | 13 [7.46 to 22] | 9.18 [5.17 to 16] | 4.78 [2.68 to 8.54] | 5.32 [3.08 to 9.19] | 1.05 [0.9 to 1.23]
  M01-0240364(NadA) - month 7 (n=44,46,44,44,50,70) | 4.46 [2.63 to 7.56] | 7.43 [4.45 to 12] | 6.03 [3.54 to 10] | 3.11 [1.81 to 5.33] | 4.29 [2.6 to 7.08] | 1.07 [0.92 to 1.25]
  M01-0240364(NadA) - month 12 (n=43,43,41,40,50,71) | 3.17 [1.77 to 5.69] | 3.77 [2.12 to 6.69] | 4.65 [2.55 to 8.47] | 2.52 [1.38 to 4.62] | 2.17 [1.26 to 3.72] | 1.03 [0.87 to 1.22]

13. Secondary Outcome: GMT Against Serogroups A, C, W, and Y at Month 0 Through Month 12 Following Vaccination at 0, 2 and 6 Months With One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean hSBA Titers Against Serogroup B Test Strains after first (month 1) and second (month 3) vaccination during the parent study NCT01210885, after 6 month of the first vaccination (6 month) in the parent study and after the third vaccination (month 7) and 6 month after the third vaccination (month 12) with One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Time Frame: At month 1, 3, 6, 7 and 12
Population: Analysis was done by MITT Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 73
Titers
  Ser. A - month 1 (n=24,24,24,25,23,70) | 42 [19 to 92] | 98 [45 to 213] | 44 [20 to 95] | 46 [21 to 98] | 4.35 [1.97 to 9.6] | 107 [66 to 172]
  Ser. A - month 3 (n=25,24,25,25,23,72) | 132 [73 to 237] | 252 [139 to 456] | 185 [103 to 333] | 153 [86 to 275] | 98 [53 to 181] | 36 [25 to 52]
  Ser. A - month 6 (n=23,24,24,25,23,69) | 14 [6.54 to 32] | 40 [19 to 86] | 32 [15 to 69] | 19 [8.99 to 41] | 4.65 [2.12 to 10] | 20 [12 to 32]
  Ser. A - month 7 (n=24,24,21,25,22,71) | 247 [124 to 495] | 296 [149 to 591] | 253 [121 to 530] | 256 [130 to 503] | 140 [68 to 289] | 21 [13 to 31]
  Ser. A - month 12 (n=25,23,21,25,22,71) | 33 [16 to 68] | 58 [27 to 123] | 47 [21 to 103] | 38 [18 to 78] | 11 [5.1 to 24] | 14 [9.03 to 22]
  Ser. C - month 1 (n=25,24,24,25,23,71) | 125 [68 to 230] | 87 [47 to 161] | 112 [61 to 208] | 74 [41 to 136] | 5.93 [3.16 to 11] | 75 [51 to 109]
  Ser. C - month 3 (n=25,24,25,24,23,71) | 482 [318 to 731] | 384 [252 to 585] | 346 [228 to 523] | 381 [250 to 580] | 20 [13 to 31] | 45 [35 to 58]
  Ser. C - month 6 (n=22,24,24,24,21,70) | 182 [111 to 297] | 143 [90 to 229] | 157 [98 to 251] | 118 [74 to 189] | 4.58 [2.77 to 7.57] | 23 [17 to 31]
  Ser. C - month 7 (n=23,24,23,25,22,72) | 676 [410 to 1114] | 676 [416 to 1097] | 636 [387 to 1046] | 553 [344 to 891] | 33 [20 to 55] | 18 [13 to 24]
  Ser. C - month 12 (n=25,23,21,25,23,72) | 202 [123 to 334] | 185 [110 to 309] | 153 [89 to 263] | 157 [96 to 258] | 7.8 [4.65 to 13] | 14 [10 to 19]
  Ser. W - month 1 (n=25,24,24,25,23,72) | 152 [92 to 253] | 180 [108 to 300] | 237 [141 to 396] | 144 [87 to 238] | 19 [11 to 32] | 210 [154 to 287]
  Ser. W - month 3 (n=25,24,25,24,23,72) | 398 [285 to 557] | 455 [324 to 639] | 499 [357 to 697] | 406 [289 to 570] | 139 [98 to 197] | 166 [135 to 204]
  Ser. W - month 6 (n=24,24,25,24,22,69) | 166 [105 to 261] | 176 [112 to 275] | 191 [123 to 297] | 148 [94 to 231] | 10 [6.28 to 16] | 117 [88 to 154]
  Ser. W - month 7 (n=23,24,21,25,21,72) | 640 [405 to 1014] | 670 [432 to 1039] | 876 [548 to 1402] | 627 [407 to 965] | 116 [72 to 187] | 121 [93 to 159]
  Ser. W - month 12(n=24,22,19,24,23,69) | 264 [159 to 438] | 258 [153 to 433] | 257 [147 to 449] | 212 [128 to 349] | 17 [10 to 29] | 75 [55 to 103]
  Ser. Y - month 1 (n=25,24,23,25,23,73) | 75 [44 to 129] | 48 [28 to 82] | 62 [36 to 109] | 71 [42 to 121] | 4.38 [2.51 to 7.67] | 92 [66 to 128]
  Ser. Y - month 3 (n=25,24,25,25,23,73) | 225 [154 to 328] | 179 [122 to 262] | 214 [147 to 312] | 170 [117 to 247] | 4.91 [3.32 to 7.26] | 72 [57 to 91]
  Ser. Y - month 6 (n=24,24,24,25,23,72) | 185 [102 to 336] | 216 [119 to 390] | 147 [81 to 267] | 121 [68 to 216] | 1.69 [0.92 to 3.09] | 84 [58 to 120]
  Ser. Y - month 7 (n=25,24,24,25,22,72) | 648 [362 to 1162] | 590 [327 to 1066] | 599 [331 to 1085] | 408 [229 to 728] | 2.56 [1.38 to 4.77] | 75 [52 to 108]
  Ser. Y - month 12 (n=25,23,21,25,23,70) | 295 [158 to 550] | 351 [184 to 670] | 210 [107 to 413] | 205 [110 to 381] | 1.46 [0.76 to 2.78] | 47 [31 to 69]

14. Secondary Outcome: GMR Against Serogroups A, C, W, and Y at Month 0 Through Month 12 Following Vaccination at 0, 2 and 6 Months With One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Description: Antibody response was measured as Geometric Mean Ratios (95%CI) Against Serogroup B Test Strains after first (month 1) and second (month 3) vaccination during the parent study NCT01210885, after 6 month of the first vaccination (6 month) in the parent study and after the third vaccination (month 7) and 6 month after the third vaccination (month 12) with One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Time Frame: At month 1, 3, 6, 7 and 12
Population: Analysis was done by MITT Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 73
Ratio
  Ser. A - month 1 (n=24,24,24,25,23,70) | 32 [15 to 71] | 71 [32 to 155] | 35 [16 to 77] | 33 [15 to 72] | 3.45 [1.54 to 7.73] | 78 [48 to 127]
  Ser. A - month 3 (n=25,24,25,25,23,72) | 99 [53 to 185] | 176 [94 to 330] | 150 [81 to 280] | 109 [59 to 202] | 79 [42 to 150] | 26 [18 to 38]
  Ser. A - month 6 (n=23,24,24,25,23,69) | 11 [4.86 to 24] | 29 [13 to 63] | 25 [12 to 56] | 14 [6.47 to 30] | 3.69 [1.66 to 8.2] | 15 [9.12 to 24]
  Ser. A - month 7 (n=24,24,21,25,22,71) | 190 [94 to 385] | 214 [106 to 432] | 201 [95 to 425] | 187 [94 to 372] | 110 [53 to 230] | 15 [9.87 to 23]
  Ser. A - month 12 (n=25,23,21,25,22,71) | 25 [12 to 52] | 42 [20 to 90] | 36 [16 to 81] | 28 [13 to 57] | 8.75 [4.01 to 19] | 11 [6.65 to 17]
  Ser. C - month 1 (n=25,24,24,25,23,70) | 23 [11 to 45] | 19 [9.55 to 38] | 26 [13 to 52] | 14 [7.09 to 28] | 1.51 [0.74 to 3.07] | 16 [11 to 25]
  Ser. C - month 3 (n=25,24,25,24,23,70) | 80 [44 to 143] | 81 [45 to 148] | 75 [42 to 135] | 63 [35 to 114] | 5.17 [2.81 to 9.52] | 9.54 [6.61 to 14]
  Ser. C - month 6 (n=22,24,24,24,21,69) | 33 [18 to 61] | 31 [17 to 56] | 33 [19 to 60] | 22 [12 to 39] | 1.16 [0.62 to 2.18] | 5.14 [3.57 to 7.39]
  Ser. C - month 7 (n=23,24,23,25,22,71) | 115 [62 to 214] | 146 [80 to 266] | 139 [75 to 258] | 100 [56 to 181] | 9.09 [4.84 to 17] | 3.9 [2.7 to 5.64]
  Ser. C - month 12 (n=25,23,21,25,23,71) | 37 [21 to 67] | 41 [22 to 75] | 33 [18 to 63] | 30 [17 to 53] | 2.01 [1.09 to 3.69] | 3.06 [2.12 to 4.4]
  Ser. W - month 1 (n=25,24,24,25,23,72) | 6.44 [3.12 to 13] | 9.65 [4.64 to 20] | 13 [6.09 to 27] | 6.3 [3.07 to 13] | 0.81 [0.38 to 1.72] | 10 [6.49 to 16]
  Ser. W - month 3 (n=25,24,25,24,23,72) | 15 [6.85 to 33] | 24 [11 to 52] | 24 [11 to 53] | 14 [6.51 to 31] | 5.42 [2.42 to 12] | 7.32 [4.53 to 12]
  Ser. W - month 6 (n=24,24,25,24,22,69) | 6.45 [3.03 to 14] | 9.27 [4.4 to 20] | 9.6 [4.6 to 20] | 6.36 [3.02 to 13] | 0.45 [0.21 to 0.98] | 5.17 [3.25 to 8.24]
  Ser. W - month 7 (n=23,24,21,25,21,72) | 24 [11 to 54] | 35 [16 to 76] | 41 [18 to 94] | 26 [12 to 55] | 4.78 [2.08 to 11] | 5.47 [3.4 to 8.8]
  Ser. W - month 12 (n=24,22,19,24,23,69) | 11 [4.99 to 24] | 15 [6.76 to 34] | 15 [6.38 to 37] | 9.44 [4.32 to 21] | 0.75 [0.34 to 1.67] | 3.62 [2.21 to 5.94]
  Ser. Y - month 1 (n=25,24,23,25,23,73) | 15 [8.32 to 28] | 9.78 [5.33 to 18] | 13 [6.88 to 24] | 15 [8.2 to 27] | 1.02 [0.55 to 1.9] | 16 [11 to 23]
  Ser. Y - month 3 (n=25,24,25,25,23,73) | 43 [26 to 71] | 35 [21 to 58] | 43 [26 to 72] | 34 [21 to 56] | 1.13 [0.67 to 1.9] | 12 [8.54 to 16]
  Ser. Y - month 6 (n=24,24,24,25,23,72) | 36 [18 to 70] | 43 [22 to 84] | 30 [15 to 59] | 25 [13 to 48] | 0.39 [0.2 to 0.78] | 14 [9.04 to 21]
  Ser. Y - month 7 (n=25,24,24,25,22,72) | 123 [63 to 242] | 115 [58 to 227] | 129 [65 to 257] | 81 [42 to 159] | 0.55 [0.27 to 1.14] | 12 [7.76 to 18]
  Ser. Y - month 12 (n=25,23,21,25,23,70) | 56 [28 to 114] | 67 [32 to 139] | 43 [20 to 93] | 41 [20 to 83] | 0.33 [0.16 to 0.69] | 7.27 [4.68 to 11]

15. Secondary Outcome: GMT Against Serogroup B Test Strains at Month 0 Through Month 12 Following Vaccination at Month 0, 2 and 6 With One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Description: as for outcome 13
Time Frame: At month 1, 3, 6, 7 and 12
Population: Analysis was done by MITT Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 73
Titers
  H44/76 (fHbp) - month 1 (n=25,24,24,24,23,73) | 4.84 [2.52 to 9.3] | 14 [7 to 26] | 22 [11 to 42] | 11 [5.83 to 22] | 5.03 [2.55 to 9.9] | 1.51 [1.19 to 1.92]
  H44/76 (fHbp) - month 3 (n=25,24,24,25,23,72) | 62 [40 to 97] | 115 [73 to 180] | 153 [97 to 241] | 110 [71 to 171] | 71 [45 to 112] | 1.27 [1.07 to 1.5]
  H44/76 (fHbp) - month 6 (n=25,24,25,24,23,72) | 5.75 [3.15 to 11] | 6.56 [3.56 to 12] | 11 [5.95 to 20] | 5.41 [2.93 to 9.98] | 6.1 [3.27 to 11] | 1.18 [1.01 to 1.37]
  H44/76 (fHbp) - month 7 (n=25,24,24,25,22,73) | 108 [61 to 190] | 149 [84 to 264] | 169 [95 to 302] | 118 [67 to 208] | 104 [57 to 191] | 1.21 [1.04 to 1.4]
  H44/76 (fHbp) - month 12 (n=25,23,21,25,23,71) | 5.42 [3.22 to 9.11] | 9.63 [5.64 to 16] | 22 [12 to 38] | 8.09 [4.84 to 14] | 9.02 [5.26 to 15] | 1.13 [1 to 1.29]
  5/99 (NadA) - month 1 (n=25,24,24,25,23,72) | 54 [31 to 93] | 128 [74 to 222] | 29 [17 to 51] | 42 [24 to 71] | 157 [90 to 276] | 2.27 [1.82 to 2.85]
  5/99 (NadA) - month 3 (n=24,24,25,24,23,71) | 328 [237 to 455] | 426 [308 to 589] | 367 [267 to 506] | 382 [277 to 528] | 454 [326 to 632] | 2.11 [1.65 to 2.7]
  5/99 (NadA) - month 6 (n=25,24,24,25,23,72) | 75 [50 to 112] | 122 [81 to 183] | 48 [32 to 72] | 84 [56 to 125] | 156 [103 to 237] | 1.74 [1.36 to 2.22]
  5/99 (NadA) - month 7 (n=25,24,24,25,23,73) | 530 [361 to 779] | 741 [502 to 1092] | 674 [456 to 996] | 527 [360 to 771] | 856 [575 to 1274] | 1.93 [1.5 to 2.48]
  5/99 (NadA) - month 12 (n=25,23,21,25,23,72) | 140 [89 to 220] | 202 [127 to 322] | 126 [77 to 206] | 127 [81 to 199] | 274 [172 to 439] | 1.53 [1.25 to 1.88]
  NZ98/254 (PorA) - month 1 (n=25,24,24,25,23,72) | 2.13 [1.41 to 3.21] | 2.22 [1.46 to 3.36] | 6.22 [4.09 to 9.45] | 2.92 [1.95 to 4.39] | 1.76 [1.15 to 2.7] | 1.51 [1.32 to 1.74]
  NZ98/254 (PorA) - month 3 (n=25,24,25,24,23,72) | 2.87 [1.87 to 4.4] | 3.14 [2.04 to 4.83] | 18 [12 to 27] | 8.95 [5.85 to 14] | 2.75 [1.77 to 4.28] | 1.49 [1.29 to 1.72]
  NZ98/254 (PorA) - month 6 (n=25,24,24,25,23,72) | 1.9 [1.29 to 2.81] | 1.85 [1.25 to 2.74] | 3.33 [2.24 to 4.96] | 1.83 [1.24 to 2.69] | 1.83 [1.22 to 2.73] | 1.15 [1.05 to 1.25]
  NZ98/254 (PorA) - month 7 (n=25,24,24,25,23,73) | 2.3 [1.49 to 3.54] | 3.24 [2.09 to 5.02] | 23 [15 to 35] | 12 [7.5 to 18] | 2.65 [1.69 to 4.14] | 1.2 [1.07 to 1.33]
  NZ98/254 (PorA) - month 12 (n=25,23,21,25,23,72) | 1.41 [0.98 to 2.02] | 1.94 [1.34 to 2.81] | 5.01 [3.4 to 7.39] | 2.39 [1.68 to 3.42] | 1.79 [1.23 to 2.59] | 1.15 [1.05 to 1.25]
  M14459 (fHBP) - month 1 (n=25,24,24,25,23,72) | 1.87 [1.2 to 2.91] | 2.78 [1.78 to 4.36] | 4.4 [2.8 to 6.91] | 2.69 [1.69 to 4.29] | 2.08 [1.32 to 3.3] | 1.26 [1.08 to 1.47]
  M14459 (fHBP) - month 3 (n=25,24,25,24,23,70) | 5.94 [3.47 to 10] | 15 [8.59 to 25] | 22 [13 to 38] | 11 [6.03 to 19] | 9.66 [5.55 to 17] | 1.29 [1.1 to 1.51]
  M14459 (fHBP) - month 6 (n=25,24,25,25,23,71) | 2.25 [1.54 to 3.3] | 2.64 [1.8 to 3.89] | 4 [2.73 to 5.86] | 2.11 [1.42 to 3.15] | 2.27 [1.53 to 3.37] | 1.28 [1.11 to 1.49]
  M14459 (fHBP) - month 7 (n=25,24,23,25,22,73) | 14 [9.12 to 22] | 23 [14 to 36] | 41 [26 to 65] | 17 [11 to 27] | 11 [6.77 to 17] | 1.28 [1.1 to 1.49]
  M14459 (fHBP) - month 12 (n=25,23,21,25,23,72) | 1.79 [1.25 to 2.57] | 2.63 [1.81 to 3.81] | 5.99 [4.06 to 8.85] | 2.35 [1.61 to 3.43] | 2.8 [1.93 to 4.07] | 1.37 [1.15 to 1.64]
  M07-0241084(NHBA) - month 1 (n=25,24,23,23,23,72) | 3.42 [2.33 to 5.02] | 3.23 [2.19 to 4.75] | 6.8 [4.57 to 10] | 5.73 [3.76 to 8.71] | 4.07 [2.76 to 6.01] | 2.68 [1.93 to 3.7]
  M07-0241084 (NHBA) - month 3 (n=25,24,22,21,22,68) | 4.04 [2.75 to 5.93] | 5.1 [3.46 to 7.53] | 12 [8.04 to 19] | 8.09 [5.18 to 13] | 6.48 [4.35 to 9.66] | 2.85 [2.08 to 3.91]
  M07-0241084 (NHBA) - month 6 (n=25,23,23,25,23,70) | 3.27 [2.26 to 4.73] | 3.21 [2.19 to 4.69] | 5.91 [3.99 to 8.74] | 4.57 [3.08 to 6.78] | 3.67 [2.52 to 5.34] | 2.99 [2.16 to 4.14]
  M07-0241084 (NHBA) - month 7 (n=25,23,22,25,21,72) | 12 [7.85 to 19] | 8.91 [5.64 to 14] | 33 [20 to 53] | 22 [14 to 35] | 11 [6.65 to 17] | 3.03 [2.22 to 4.15]
  M07-0241084(NHBA) - month 12 (n=25,23,21,25,23,70) | 2.77 [1.85 to 4.13] | 3.05 [2.01 to 4.61] | 9.99 [6.39 to 16] | 4.92 [3.2 to 7.56] | 5.74 [3.82 to 8.64] | 2.91 [2.06 to 4.12]
  M01-0240364 (NadA) - month 1 (n=23,24,24,25,23,72) | 2.94 [1.32 to 6.58] | 10 [4.75 to 22] | 6 [2.71 to 13] | 5.52 [2.46 to 12] | 3.84 [1.74 to 8.52] | 1.12 [0.98 to 1.29]
  M01-0240364 (NadA) - month 3 (n=25,24,24,24,23,70) | 41 [19 to 88] | 245 [113 to 532] | 126 [57 to 280] | 205 [91 to 459] | 226 [102 to 501] | 1.41 [1.07 to 1.85]
  M01-0240364 (NadA) - month 6 (n=25,21,24,24,21,71) | 4.39 [2.09 to 9.19] | 9.54 [4.3 to 21] | 7.3 [3.44 to 15] | 9.08 [4.1 to 20] | 7.87 [3.54 to 18] | 1.18 [1 to 1.39]
  M01-0240364 (NadA) - month 7 (n=24,23,24,25,23,71) | 294 [147 to 589] | 513 [255 to 1035] | 409 [202 to 829] | 280 [137 to 572] | 507 [251 to 1027] | 1.18 [1 to 1.39]
  M01-0240364(NadA) - month 12 (n=23,21,20,25,22,72) | 7.32 [3.4 to 16] | 24 [11 to 54] | 17 [7.37 to 38] | 19 [8.71 to 41] | 41 [19 to 88] | 1.15 [0.97 to 1.37]

16. Secondary Outcome: GMR Against Serogroup B Test Strains at Month 0 Through Month 12 Following Vaccination at Month 0, 2 and 6 With One of Four MenABCWY Formulations, rMenB, or MenACWY/Placebo
Description: as for outcome 14
Time Frame: At month 1, 3, 6, 7 and 12
Population: Analysis was done by MITT Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 3ABCWY | 3ABx2CWY | 3ABCWY+OMV | 3ABCWYqOMV | 3 B | 1ACWY
Number analyzed (Participants) | 25 | 24 | 25 | 25 | 23 | 73
Ratio
  H44/76 (fHbp) - month 1 (n=25,24,24,24,23,73) | 3.79 [1.97 to 7.29] | 11 [5.45 to 20] | 17 [8.59 to 33] | 8.95 [4.62 to 17] | 3.92 [1.99 to 7.72] | 1.15 [0.98 to 1.35]
  H44/76 (fHbp) - month 3 (n=25,24,24,25,23,72) | 48 [29 to 78] | 86 [52 to 143] | 111 [67 to 185] | 90 [55 to 147] | 53 [32 to 89] | 1.05 [0.89 to 1.24]
  H44/76 (fHbp) - month 6 (n=25,24,25,24,23,72) | 4.47 [2.43 to 8.23] | 5.06 [2.73 to 9.37] | 8.28 [4.5 to 15] | 4.31 [2.32 to 8.01] | 4.7 [2.5 to 8.85] | 0.89 [0.78 to 1.02]
  H44/76 (fHbp) - month 7 (n=25,24,24,25,22,73) | 83 [46 to 150] | 113 [63 to 206] | 126 [69 to 229] | 95 [53 to 170] | 79 [42 to 147] | 0.92 [0.79 to 1.06]
  H44/76 (fHbp) - month 12 (n=25,23,21,25,23,71) | 4.22 [2.49 to 7.14] | 7.44 [4.33 to 13] | 16 [9.28 to 29] | 6.45 [3.83 to 11] | 6.97 [4.04 to 12] | 0.86 [0.73 to 1.01]
  5/99 (NadA) - month 1 (n=25,24,24,25,23,72) | 23 [12 to 42] | 60 [32 to 110] | 14 [7.59 to 26] | 19 [11 to 35] | 79 [42 to 148] | 1 [0.85 to 1.18]
  5/99 (NadA) - month 3 (n=24,24,25,24,23,71) | 131 [79 to 216] | 197 [120 to 324] | 182 [112 to 298] | 182 [111 to 299] | 233 [140 to 387] | 1 [0.8 to 1.26]
  5/99 (NadA) - month 6 (n=25,24,24,25,23,72) | 31 [19 to 53] | 56 [34 to 95] | 24 [14 to 41] | 39 [23 to 64] | 79 [46 to 134] | 0.78 [0.61 to 0.99]
  5/99 (NadA) - month 7 (n=25,24,24,25,23,73) | 221 [133 to 368] | 344 [206 to 574] | 325 [194 to 545] | 244 [147 to 403] | 435 [257 to 736] | 0.86 [0.68 to 1.08]
  5/99 (NadA) - month 12 (n=25,23,21,25,23,72) | 58 [34 to 101] | 95 [54 to 167] | 62 [34 to 111] | 58 [34 to 100] | 138 [78 to 243] | 0.7 [0.59 to 0.83]
  NZ98/254 (PorA) - month 1 (n=25,24,24,25,23,72) | 1.25 [0.82 to 1.9] | 1.32 [0.86 to 2.02] | 3.63 [2.37 to 5.57] | 1.71 [1.13 to 2.6] | 1.06 [0.68 to 1.63] | 1 [0.87 to 1.16]
  NZ98/254 (PorA) - month 3 (n=25,24,25,24,23,72) | 1.67 [1.07 to 2.6] | 1.86 [1.19 to 2.91] | 10 [6.67 to 16] | 5.16 [3.31 to 8.06] | 1.64 [1.04 to 2.6] | 0.99 [0.83 to 1.17]
  NZ98/254 (PorA) - month 6 (n=25,24,24,25,23,72) | 1.11 [0.73 to 1.67] | 1.1 [0.73 to 1.67] | 1.93 [1.27 to 2.92] | 1.06 [0.71 to 1.59] | 1.09 [0.71 to 1.67] | 0.76 [0.65 to 0.89]
  NZ98/254 (PorA) - month 7 (n=25,24,24,25,23,73) | 1.33 [0.84 to 2.1] | 1.93 [1.21 to 3.07] | 13 [8.14 to 21] | 6.66 [4.23 to 10] | 1.59 [0.99 to 2.55] | 0.8 [0.67 to 0.94]
  NZ98/254 (PorA) - month 12 (n=25,23,21,25,23,72) | 0.81 [0.55 to 1.19] | 1.13 [0.76 to 1.69] | 2.81 [1.85 to 4.27] | 1.37 [0.94 to 2.02] | 1.06 [0.71 to 1.58] | 0.77 [0.66 to 0.9]
  M14459 (fHBP) - month 1 (n=25,24,24,22,23,71) | 1.46 [0.94 to 2.27] | 2.18 [1.39 to 3.4] | 3.46 [2.2 to 5.42] | 2.12 [1.33 to 3.38] | 1.64 [1.04 to 2.59] | 0.95 [0.87 to 1.03]
  M14459 (fHBP) - month 3 (n=25,24,25,22,23,69) | 4.41 [2.57 to 7.57] | 11 [6.28 to 19] | 17 [9.77 to 29] | 8.26 [4.68 to 15] | 7.4 [4.22 to 13] | 1.04 [0.9 to 1.2]
  M14459 (fHBP) - month 6 (n=25,24,25,22,23,70) | 1.73 [1.18 to 2.53] | 2.02 [1.37 to 2.96] | 3.1 [2.12 to 4.54] | 1.66 [1.11 to 2.48] | 1.77 [1.19 to 2.63] | 0.99 [0.87 to 1.12]
  M14459 (fHBP) - month 7 (n=25,24,23,22,22,72) | 10 [6.66 to 16] | 16 [10 to 26] | 31 [19 to 49] | 13 [8.26 to 21] | 8.18 [5.06 to 13] | 0.97 [0.83 to 1.13]
  M14459 (fHBP) - month 12 (n=25,23,21,22,23,71) | 1.35 [0.94 to 1.94] | 1.97 [1.35 to 2.86] | 4.57 [3.09 to 6.77] | 1.83 [1.25 to 2.68] | 2.16 [1.48 to 3.14] | 1.03 [0.87 to 1.24]
  M07-0241084 (NHBA) - month 1 (n=24,23,22,20,23,66) | 1.28 [0.87 to 1.89] | 1.19 [0.8 to 1.75] | 2.5 [1.67 to 3.74] | 2.1 [1.38 to 3.21] | 1.55 [1.05 to 2.29] | 1.02 [0.87 to 1.19]
  M07-0241084 (NHBA) - month 3 (n=24,23,20,18,22,65) | 1.52 [1 to 2.3] | 1.82 [1.2 to 2.77] | 4.54 [2.89 to 7.11] | 2.81 [1.74 to 4.54] | 2.56 [1.67 to 3.93] | 1.13 [0.89 to 1.44]
  M07-0241084 (NHBA) - month 6 (n=24,22,21,21,23,65) | 1.22 [0.83 to 1.8] | 1.14 [0.76 to 1.7] | 2.14 [1.42 to 3.23] | 1.62 [1.07 to 2.46] | 1.42 [0.95 to 2.1] | 1.2 [0.97 to 1.49]
  M07-0241084 (NHBA) - month 7 (n=24,22,20,21,21,66) | 4.55 [2.84 to 7.29] | 3.1 [1.9 to 5.05] | 12 [6.98 to 20] | 7.7 [4.65 to 13] | 4.15 [2.49 to 6.9] | 1.21 [0.96 to 1.51]
  M07-0241084 (NHBA) - month 12(n=24,22,19,21,23,64) | 1.03 [0.67 to 1.59] | 1.07 [0.68 to 1.66] | 3.56 [2.21 to 5.75] | 1.73 [1.09 to 2.74] | 2.24 [1.44 to 3.46] | 1.19 [0.9 to 1.58]
  M01-0240364 (NadA) - month 1 (n=23,24,23,22,23,71) | 2.33 [1.04 to 5.2] | 8.23 [3.79 to 18] | 4.84 [2.19 to 11] | 4.48 [2 to 10] | 3.12 [1.41 to 6.91] | 1 [0.86 to 1.16]
  M01-0240364 (NadA) - month 3 (n=25,24,23,22,23,69) | 31 [14 to 68] | 190 [85 to 424] | 105 [46 to 239] | 177 [77 to 408] | 196 [86 to 446] | 1.28 [1.01 to 1.63]
  M01-0240364 (NadA) - month 6 (n=25,21,24,21,21,70) | 3.41 [1.62 to 7.2] | 7.46 [3.33 to 17] | 5.97 [2.79 to 13] | 7.56 [3.39 to 17] | 6.57 [2.93 to 15] | 1.05 [0.9 to 1.23]
  M01-0240364 (NadA) - month 7 (n=24,23,23,22,23,70) | 226 [111 to 459] | 401 [196 to 820] | 336 [164 to 690] | 236 [114 to 488] | 428 [209 to 879] | 1.07 [0.92 to 1.25]
  M01-0240364 (NadA) - month 12(n=23,21,20,22,22,71) | 5.61 [2.58 to 12] | 19 [8.45 to 42] | 14 [6.13 to 32] | 16 [7.28 to 35] | 34 [16 to 76] | 1.03 [0.87 to 1.22]

17. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Vaccination
Description: Unsolicited AEs were collected with onset from Day 1 through Day 7 After Vaccination. One subject initially randomized to group 3ABCWYqOMV and supposed to receive rMenB+1/4OMV+ACWY as the third vaccination, actually received Tdap as the third vaccination and was included in 2ABCWYqOMV group for the safety analysis.
Time Frame: From Day 1 to Day 7 after vaccination
Population: Analysis was done on the Safety Set (all subjects in the exposed set who provided post-vaccination unsolicited AE data).
Measure: Number; unit: Number of Subjects
Arm/Group | 3ABCWY | 2ABCWY | 3ABx2CWY | 2ABx2CWY | 3ABCWY+OMV | 2ABCWY+OMV | 3ABCWYqOMV | 2ABCWYqOMV | 3 B | 2 B | 1ACWY
Number analyzed (Participants) | 24 | 49 | 24 | 49 | 25 | 48 | 24 | 50 | 23 | 50 | 73
Number of Subjects
  Any AEs | 3 | 6 | 1 | 4 | 2 | 3 | 3 | 2 | 2 | 6 | 6
  At least possibly related AEs | 1 | 4 | 0 | 2 | 1 | 1 | 3 | 0 | 1 | 3 | 3
  Serious AEs | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  At least possibly related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

18. Secondary Outcome: Numbers of Subjects With Other Unsolicited AEs
Description: Unsolicited AEs were collected from Day 8 After vaccination Through Study Termination. One subject initially randomized to group 3ABCWYqOMV and supposed to receive rMenB+1/4OMV+ACWY as the third vaccination, actually received Tdap as the third vaccination and was included in 2ABCWYqOMV group for the safety analysis.
Time Frame: Day 8 After vaccination Through Study Termination, up to 6 months
Population: Analysis was done on the Safety Set (all subjects in the exposed set who provided post-vaccination unsolicited AE data).
Measure: Number; unit: Number of Subjects
Arm/Group | 3ABCWY | 2ABCWY | 3ABx2CWY | 2ABx2CWY | 3ABCWY+OMV | 2ABCWY+OMV | 3ABCWYqOMV | 2ABCWYqOMV | 3 B | 2 B | 1ACWY
Number analyzed (Participants) | 24 | 48 | 24 | 49 | 25 | 48 | 24 | 50 | 23 | 50 | 73
Number of Subjects
  Medically attended AEs | 5 | 7 | 4 | 10 | 6 | 7 | 2 | 5 | 4 | 14 | 15
  AEs leading to Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least possibly related AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  SAEs | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  At least possibly related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events (AEs) After Vaccination
Description: Solicited local and systemic AEs were collected daily for 7 days (day 1 through day 7) after vaccination. One subject initially randomized to group 3ABCWYqOMV and supposed to receive rMenB+1/4OMV+ACWY as the third vaccination, actually received Tdap as the third vaccination and was included in 2ABCWYqOMV group for the safety analysis.
Time Frame: From Day 1 to Day 7 after vaccination
Population: Analysis was done on Safety Set (all subjects in the exposed set who provided post-vaccination solicited AE data).
Measure: Number; unit: Number of Subjects
Arm/Group | 3ABCWY | 2ABCWY | 3ABx2CWY | 2ABx2CWY | 3ABCWY+OMV | 2ABCWY+OMV | 3ABCWYqOMV | 2ABCWYqOMV | 3 B | 2 B | 1ACWY
Number analyzed (Participants) | 24 | 48 | 24 | 49 | 25 | 48 | 24 | 50 | 23 | 50 | 73
Number of Subjects
  Any Solicited Local AEs | 18 | 33 | 18 | 35 | 23 | 36 | 20 | 30 | 17 | 38 | 53
  Injection site erythema | 5 | 13 | 7 | 12 | 12 | 11 | 13 | 3 | 9 | 13 | 19
  Injection site induration | 7 | 14 | 11 | 12 | 10 | 17 | 11 | 6 | 7 | 14 | 18
  Injection site pain | 18 | 33 | 15 | 35 | 23 | 35 | 19 | 30 | 17 | 36 | 52
  Swelling | 5 | 11 | 9 | 10 | 10 | 14 | 13 | 5 | 7 | 14 | 14
  Any Solicited Systemic AEs | 10 | 33 | 14 | 25 | 20 | 23 | 18 | 24 | 14 | 34 | 43
  Chills | 3 | 10 | 4 | 2 | 7 | 7 | 4 | 5 | 5 | 5 | 8
  Malaise | 6 | 12 | 7 | 14 | 8 | 9 | 7 | 8 | 5 | 13 | 13
  Myalgia | 6 | 23 | 9 | 20 | 15 | 18 | 14 | 19 | 9 | 21 | 32
  Arthralgia | 2 | 6 | 5 | 7 | 6 | 5 | 8 | 3 | 2 | 8 | 9
  Headache | 5 | 20 | 6 | 17 | 9 | 11 | 10 | 15 | 6 | 18 | 27
  Fatigue | 3 | 9 | 3 | 9 | 5 | 11 | 4 | 7 | 3 | 10 | 9
  Nausea | 4 | 6 | 2 | 3 | 4 | 6 | 6 | 3 | 2 | 4 | 6
  Rash | 1 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2
  Fever (≥38°C) | 3 | 5 | 0 | 3 | 3 | 0 | 3 | 1 | 2 | 2 | 4
  Any other indicators of reactogenicity | 4 | 8 | 3 | 5 | 6 | 3 | 7 | 4 | 3 | 5 | 11
  Stay home | 0 | 5 | 0 | 2 | 1 | 0 | 3 | 1 | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: Safety was assessed up to 6 months after vaccination. Solicited local AEs and systemic AEs were collected daily for 7 days (day 1 through day 7) after vaccination. All unsolicited AEs including SAEs were collected for 7 days after the vaccination.
Description: The analyses for serious unsolicited adverse events (SAEs) and adverse events (AEs) were done on the safety population. One subject initially randomized to group 3ABCWYqOMV and supposed to receive rMenB+1/4OMV+ACWY as the third vaccination, actually received Tdap as the third vaccination and was included in 2ABCWYqOMV group for the safety analysis.
Arm/Group | 3ABCWY | 2ABCWY | 3ABx2CWY | 2ABx2CWY | 3ABCWY+OMV | 2ABCWY+OMV | 3ABCWYqOMV | 2ABCWYqOMV | 3 B | 2 B | 1ACWY
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/49 | 1/24 | 1/49 | 0/25 | 0/48 | 1/24 | 1/50 | 0/23 | 1/50 | 0/73
Other Adverse Events (participants affected / at risk) | 20/24 | 38/49 | 20/24 | 36/49 | 23/25 | 37/48 | 22/24 | 38/50 | 19/23 | 40/50 | 56/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3ABCWY (N=24) | 2ABCWY (N=49) | 3ABx2CWY (N=24) | 2ABx2CWY (N=49) | 3ABCWY+OMV (N=25) | 2ABCWY+OMV (N=48) | 3ABCWYqOMV (N=24) | 2ABCWYqOMV (N=50) | 3 B (N=23) | 2 B (N=50) | 1ACWY (N=73)
Appendiceal Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonsillar Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns Second Degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaccination Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3ABCWY (N=24) | 2ABCWY (N=49) | 3ABx2CWY (N=24) | 2ABx2CWY (N=49) | 3ABCWY+OMV (N=25) | 2ABCWY+OMV (N=48) | 3ABCWYqOMV (N=24) | 2ABCWYqOMV (N=50) | 3 B (N=23) | 2 B (N=50) | 1ACWY (N=73)
Nausea (Gastrointestinal disorders) | 4 | 6 | 2 | 3 | 4 | 7 | 6 | 3 | 2 | 4 | 6
Chills (General disorders) | 3 | 10 | 4 | 2 | 7 | 8 | 4 | 5 | 5 | 5 | 8
Fatigue (General disorders) | 3 | 9 | 3 | 9 | 5 | 11 | 4 | 7 | 3 | 10 | 9
Injection Site Erythema (General disorders) | 5 | 16 | 7 | 14 | 13 | 12 | 16 | 5 | 10 | 14 | 20
Injection Site Induration (General disorders) | 7 | 16 | 11 | 13 | 12 | 17 | 13 | 8 | 8 | 15 | 19
Injection Site Pain (General disorders) | 18 | 33 | 15 | 35 | 23 | 35 | 19 | 31 | 17 | 36 | 52
Injection Site Swelling (General disorders) | 5 | 11 | 9 | 11 | 11 | 14 | 14 | 6 | 8 | 14 | 16
Malaise (General disorders) | 6 | 12 | 7 | 14 | 8 | 9 | 8 | 8 | 5 | 13 | 13
Pyrexia (General disorders) | 3 | 6 | 0 | 3 | 3 | 0 | 5 | 1 | 2 | 3 | 4
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0 | 4 | 1 | 1 | 1 | 2 | 1 | 3 | 4
Athralgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 5 | 7 | 6 | 5 | 8 | 3 | 2 | 8 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 23 | 9 | 20 | 15 | 18 | 14 | 19 | 9 | 21 | 32
Headache (Nervous system disorders) | 5 | 20 | 6 | 17 | 9 | 11 | 10 | 15 | 7 | 18 | 27
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.